CLINICAL TRIAL: NCT04627701
Title: Evaluation of the Safety and Efficacy of the Omega System for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Omega Study: Evaluation of the Safety and Efficacy of the Omega System for the Treatment of BPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProArc Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-CP-20
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-05

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omega Device (Experimental)
  Interventions: Device: Omega

INTERVENTIONS:
Device: Omega — Omega Implantation

SUMMARY:
The ProArc Medical Omega system is a prostatic reshaping device that is designed to treat Lower Urinary Tract Symptoms (LUTS) due to BPH. During the procedure an implant is delivered into the prostate tissue obstructing the urethra and restricting urine flow. The delivery system uses a static diathermy incision mechanism to make a circumferential incision in the tissue surrounding the prostatic urethra into which the Omega shaped permanent implant is placed. The implant expands the obstructed area, reducing the fluid obstruction through the prostatic urethra.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥50 years of age
2. Diagnosed with symptomatic benign prostatic hyperplasia (BPH).
3. International Prostate Symptom Score (IPSS) >13.
4. Peak flow rate ≤ 12 ml/sec (with voided volume ≥ 125ml).
5. Participant understands and is willing to the informed consent form.
6. Prostate Volume between 30cc and 80cc.
7. Prostate length ≥3cm and ≤5cm

Exclusion Criteria:

1. Concomitant participation in another interventional study.
2. Unable to comply with the clinical protocol including all the follow-up requirements.
3. Vulnerable population such as inmates or developmentally delayed individuals.
4. Significant comorbidities which would affect study participation.
5. Diagnosed or suspected prostate cancer. If suspected, prostate cancer must be ruled out.
6. Any medical condition or treatment, which in the opinion of the investigator may interfere with the procedure, such as:

   * Use of concomitant medications (e.g., anticholinergics, antispasmodics, or antidepressants) affecting bladder function.
   * Patient with coagulopathy due to medications or congenital condition - inability to stop taking anticoagulants and/or antiplatelets for at least 3 days prior to the procedure or coumadin for at least 5 days prior to the procedure; low dose aspirin therapy not prohibited.
   * Alpha-blockers within 2 weeks of pre-treatment (baseline) evaluation.
   * Taking 5-alpha reductase inhibitors (5-ARI) within 6 months (3 months for type II 5-ARI) of pre-treatment (baseline) evaluation unless evidence of same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued throughout the study).
   * Patient is taking steroids. [Note: Patients approved for the trial who are using the above medications will continue using them after the trial, except for Alpha blockers]
7. Previous prostate surgery such as: TURP, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate.
8. Compromised renal function due to obstructive uropathy.
9. Active Urinary Tract Infection (UTI).
10. Obstructive or protruding median lobe
11. American Society of Anaesthesiologists score (ASA) > 3.
12. Known neurogenic bladder or neurological disorders that might affect bladder or function.
13. Recent myocardial infarction (less than three months).
14. Concomitant bladder stones.
15. Current gross hematuria.
16. Active or history of epididymitis within the past 3 months.
17. Presence of an artificial urinary sphincter or stent(s) in the urethra or prostate.
18. Confirmed or suspected malignancy of bladder.
19. History or presence of strictures in the anterior urethra or bladder neck contracture or detrusor muscle spasms.
20. Other Urethral conditions that may prevent insertion of Delivery Device into prostatic urethra.
21. Bacterial prostatitis within the last 12 months.
22. Previous rectal surgery, other than hemorrhoidectomy.
23. Current uncontrolled diabetes (i.e., hemoglobin A1c ≥ 9%).
24. Known allergy to nickel or titanium or stainless steel.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-07-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in urinary related symptoms as evidenced by IPSS score | 3 months

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Carmel Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
- Tauranga Urology Research Limited, Tauranga, New Zealand

IPD SHARING:
Plan to Share IPD: No